CLINICAL TRIAL: NCT01825330
Title: Effect of NeuroAD, Combined TMS Stimulation and Cognitive Training, on the Cognitive Function of Mild to Moderate Alzheimer Patients
Brief Title: Effect of NeuroAD on the Cognitive Function of Alzheimer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuronix Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NRX - US4
Record Dates: First submitted 2013-03-24; First posted 2013-04-05 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2015-10

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Alzheimer's; TMS; Cognitive Training; NeuroAD
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NeuroAD (Active Comparator): NeuroAD treatment, synchronized TMS and cognitive training stimulation
  Interventions: Device: TMS and cognitive stimulation
- Sham TMS+Cog (Sham Comparator): Sham device, has the same appearance and sound as the real device, combined with sham cognitive exercises. Patients come for the same number of sessions, delivers no real stimulation or cognitive training.
  Interventions: Device: sham

INTERVENTIONS:
Device: TMS and cognitive stimulation — Synchronized TMS and cognitive stimulation to 6 brain areas.
  Other Names: NeuroAD; NICE
  Arms: NeuroAD
Device: sham
  Arms: Sham TMS+Cog

SUMMARY:
The study tests the effect of the NeuroAD on Alzheimer patients' cognitive function. The NeuroAD uses non-invasive stimulation of both magnetic and cognitive training.

DETAILED DESCRIPTION:
The NeuroAD system is a combined system of Transcranial Magnetic Stimulation and cognitive training and is a non-invasive therapeutic system for the improvement of Alzheimer patients' cognitive function.

A potential participant will undergo screening procedures to confirm eligibility to participate in the study, followed by randomization procedure to one of the study groups - treatment or sham (placebo) Patient will attend the clinic 5 times a week for 6 weeks, approximately an hour every day for treatment/sham. The patient will be required to return to the clinic for follow-up.

Up to 150 patients will be enrolled in up to 10 clinical sites in the US and Israel.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 60-90 years
2. Patients diagnosed with mild or moderate stage of Alzheimer's Disease, according to the DSM-IV criteria.
3. MMSE score 18 to 26
4. ADAS-Cog above 17
5. Physical clearance for study participation as evaluated by the clinician.
6. Spouse, family member or professional caregiver agree and capable of taking care and be responsible for the participation of the patient in the study (answering questions regarding the patient's condition and assuming responsibility for medication)
7. Agreement to participate in approximately 14 weeks during the study.
8. Normal to near-normal vision and hearing with correction as needed (e.g. corrective lenses, hearing aid).
9. Fluent in English or Hebrew
10. Minimum of 8th grade education
11. If medicated for AD, then use of cholinesterase inhibitors, memantine or Ginko-biloba for at least 3 months and on stable dose for at least 60 days prior to screening.

Exclusion Criteria:

1. CDR 0, 0.5 or 3
2. Severe agitation
3. Mental retardation
4. Patient lacking capacity to consent to study participation
5. Unstable medical condition
6. Use of benzodiazepines or barbiturates 2 weeks prior to screening
7. Pharmacological immunosuppression
8. Participation in a clinical trial with any investigational agent within 6 months prior to study enrollment
9. History of Epileptic Seizures or Epilepsy
10. Contraindication for performing MRI scanning
11. Contraindication for receiving TMS treatment according to a TMS questionnaire
12. Pregnant women and women who have the ability to become pregnant unless they are on an acceptable method of contraception during the study.
13. Patients with depression, bipolar disorder or psychotic disorders or any other neurological or psychiatric condition (whether now or in the past), which the Investigator finds as interfering with the study
14. Alcoholism or drug addiction as defined by DSM-IV within last 5 years (addicted more than one year and or in remission less than 3 years) or severe sleep deprivation
15. Patients with metal implants in the head, (i.e. cochlear implants, implanted brain stimulators, aneurysm clips) with the exception of metal implants in mouth
16. Patients with personal history of either any clinically defined medical disorder (which the investigator finds as interfering with the study) or any clinically defined neurological/psychiatric disorder (other than AD), including (but not limited to): epilepsy, stroke, brain lesions, substance abuse, vitamin B12 deficiency, abnormal thyroid function, cerebrovascular condition, other neurodegenerative disease, head trauma, multiple sclerosis; or personal history of previous neurosurgery or head trauma that resulted in loss of consciousness.
17. Patients with any signs or symptoms of increased intracranial pressure, as determined in a neurological exam.
18. Cardiac pacemakers
19. Implanted medication pumps
20. Intracardiac lines
21. Significant heart disease
22. Currently taking medication that lower the seizure threshold.
23. Patients on which TMS Motor Threshold cannot be found.
24. Patient underwent TMS treatment in the past.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2013-10; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Efficacy | 7 weeks
  Change from Baseline to week 7 in ADAS-Cog score. ADAS-Cog: Alzheimer's Disease Assessment Scale - Cognitive

SECONDARY OUTCOMES:
Efficacy | 7 weeks
  Change from baseline to week 7 in CGI-C score. CGI-C: Clinical Global Impression of Change
Efficacy | 12 weeks
  Change from baseline to week 12 in ADAS-Cog score.

OTHER OUTCOMES:
Safety | 12 weeks
  Adverse events, including Serious Adverse Events occurring at any time during the trial and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Charlie Bernick, MD, Principal Investigator — Lou Ruvo Brain Center
Locations (10):
- United States (9):
  - Banner Sun Health Research Institute, Sun City, Arizona
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Miami Jewish Health Systems, Miami, Florida
  - Roskamp Institute Clinic, Sarasota, Florida
  - Palm Beach Neurology and Premiere Research Institute, West Palm Beach, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Cleveland Clinic Lou Ruvo Brain Center, Las Vegas, Nevada
  - NYU Langone Medical Center, New York, New York
  - Cleveland Clinic Center for Brain Health Lakewood Hospital, Cleveland, Ohio
- Assaf Harofe Medical Center, Beer Yaakov, Israel

REFERENCES:
- See also: Sponsor's website — http://www.neuronixmedical.com/